CLINICAL TRIAL: NCT01056887
Title: Copeptin in Differentiation of Polyuria and Polydipsia
Status: Completed | Type: Observational
Sponsor: University of Wuerzburg (Other)
Collaborators: Dr. Carson Liu Med Corp. (Industry)
Responsible Party: Prof. Dr. med. Bruno Allolio, FDAAA
Other Study IDs: 17121979; 33/07
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2010-11

CONDITIONS: Polyuria; Polydipsia
Keywords: diabetes insipidus; primary polydipsia; copeptin; Utility of plasma copeptin in differential diagnosis of polyuria/ polydipsia while performing a traditional deprivation test
MeSH Terms: conditions — Polyuria; Polydipsia; Diabetes Insipidus; Polydipsia, Psychogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Primary Polydip, D. insipidus

SUMMARY:
The differential diagnosis of patients with polyuria/ polydipsia is often complex, but important for the therapeutic strategy.

Challenging is in particular the clinical differentiation between patients with a partial Diabetes insipidus centralis and patients with primary polydipsia as underlying disease, because both groups are associated with similar urinary osmolalities.

The determination of plasma arginine vasopressin is unusual in this context, since measurement of AVP is not reliably.

C-terminal ProVasopressin (copeptin) is secreted stoichiometrically with AVP from the neurohypophysis, but has a longer half life in the circulation, and is thus easier to measure.

Therefore, the investigators will analyze in that study the diagnostic utility of plasma copeptin in the differential diagnosis of polyuria and polydipsia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with polydipsia/ polyuria, with indication for performing a deprivation test
* > 18 years

Exclusion Criteria:

* dDAVP during the last 14d
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy probands Patients with diabetes insipdus centralis totalis/ partials Patients with diabetes insipidus renalis Patients with primary polydipsia
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Univ Hospital Wuerzburg, Würzburg, Bavaria, Germany

REFERENCES:
- [Derived] Fenske W, Quinkler M, Lorenz D, Zopf K, Haagen U, Papassotiriou J, Pfeiffer AF, Fassnacht M, Stork S, Allolio B. Copeptin in the differential diagnosis of the polydipsia-polyuria syndrome--revisiting the direct and indirect water deprivation tests. J Clin Endocrinol Metab. 2011 May;96(5):1506-15. doi: 10.1210/jc.2010-2345. Epub 2011 Mar 2. PMID 21367924